CLINICAL TRIAL: NCT03869073
Title: Randomized, Double-blind, Placebo-controlled Phase 2a Trial of Efficacy and Safety of Evolocumab for PCSK9 Lowering in Early Acute Sepsis
Brief Title: Evolocumab for PCSK9 Lowering in Early Acute Sepsis (The PLEASe Study)
Acronym: PLEASe
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, john boyd, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H18-00917
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Sepsis
Keywords: Bacterial; Infection; Blood; Systemic; ICU
MeSH Terms: conditions — Sepsis; Infections | interventions — evolocumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Upon enrolling in the study participants will be randomized into one of three possible treatment arms: 420mg single dose at baseline, 840mg single dose at baseline, or placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low Dose (Experimental): This treatment arm will receive the highest dose of evolocumab currently marketed and approved: 420mg. The dose will be given at a single time point within 4 hours of randomization. The dose will be administered through three subcutaneous injections, each in a different quadrant of the abdomen.
  Interventions: Drug: Evolocumab
- High Dose (Experimental): This treatment arm will receive double the highest dose of evolocumab currently marketed and approved: 840mg. The dose will be given at a single time point within 4 hours of randomization. The dose will be administered through three subcutaneous injections, each in a different quadrant of the abdomen.
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): This treatment arm will receive saline solution. The dose will be given at a single time point within 4 hours of randomization. The dose will be administered through three subcutaneous injections, each in a different quadrant of the abdomen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — Three pre-filled shrouded syringes for subcutaneous injection in abdomen.
  Other Names: Repatha
  Arms: High Dose; Low Dose
Drug: Placebo — Preservative free 0.9% sodium chloride. Three pre-filled shrouded syringes for subcutaneous injection in abdomen.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study evaluates using evolocumab, a currently approved and marketed biologic drug, in a novel way. Patients who present to the emergency room or intensive care unit (ICU) with severe infection are eligible. Either the patient or their designated decision maker will be approached for consent. If they choose to participate they will be given either a single dose of evolocumab, a higher single dose of evolocumab,or a single dose of placebo. Participants will be followed during their stay in the ICU and will receive follow up phone calls at Day 28 and 90.

DETAILED DESCRIPTION:
Evolocumab is currently approved and marketed in USA and Canada for lowering cholesterol levels. Evolocumab is an anti-PSCK9 monoclonal antibody, and functions by binding PSCK9 (an inhibitor of LDL removal) and blocking its function. Evidence suggests that since evolocumab increases the removal rate of low-density lipoproteins from the body, it might also help increase the removal of bacterial components that are attached to circulating lipids during sepsis. Quickly removing these bacterial components could prevent a strong and rapid immune response that often leads to organ failure and death in sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* At least 19 years of age
* Known or suspected infection
* AND one or more of the following organ dysfunctions judged due to sepsis:

  1. Cardiovascular- refractory hypotension (a systolic blood pressure (SBP) < 90 mm Hg or mean arterial pressure (MAP) < 60 mm Hg despite an IV fluid challenge of at least 30 ml/kg fluids), or use of vasopressor(s) to maintain SAP > 90 mm Hg or MAP > 60 mm Hg, or;
  2. Respiratory: PaO2/FiO2 < 300 or PaO2/FiO2 < 200 if lung is the only organ dysfunction or SaO2:FiO2 150

Exclusion Criteria:

* Known pregnancy
* Underlying severe congestive heart failure (New York Heart Association (NYHA) IV), severe COPD (need for chronic oxygen or mechanical ventilation), severe liver disease (Child-Pugh Class C), cancer requiring chemotherapy, or transplantation (bone marrow, heart, lung, liver, pancreas, or small bowel) in the past 6 months or likely within the next 6 months
* Previous episode of sepsis during that hospital admission
* Absolute Neutrophil Count < 500/mm³
* CD4 count < 50/mm³
* Treating physician deems aggressive care unsuitable (i.e. no commitment to active care)
* Participation in another interventional drug study within previous 1 month
* Allergic to the study drug or any of its components
* Lactation
* Have signed a Do No Resuscitate (DNR) Form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-02-11 (Estimated); Study Completion 2021-02-11 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma LTA and LPS curves | 7 days or less (as data is collected from participants only while they are admitted to critical care, they may be discharged or moved to a different ward before day 7 and therefore subsequent time points would be not be collected)
  Determine whether evolocumab decreases plasma levels of bacterial LPS and LTA, at 6, 24, 48 and 72 hours, and day 7 by comparing the area under the operating curve between arms.

SECONDARY OUTCOMES:
Levels of LDL-C | 7 days or less (as data is collected from participants only while they are admitted to critical care, they may be discharged or moved to a different ward before day 7 and therefore subsequent time points would be not be collected)
  Measure levels (concentration; e.g. ug/mL) of low-density lipoprotein-cholesterol (LDL-C) at 24, 48, and 72 hours, and day 7, and compare area under the plasma cytokine curve between arms.
Levels of cytokines IL-6, TNF-alpha and IL-8 | 7 days or less (as data is collected from participants only while they are admitted to critical care, they may be discharged or moved to a different ward before day 7 and therefore subsequent time points would be not be collected)
  Measure levels (concentration; e.g. ug/mL) of cytokines (IL-6, TNF-alpha and IL-8) at 24, 48, and 72 hours, and day 7, and compare area under the plasma cytokine curve between arms.
Concentration of circulating evolocumab and circulating free PCSK9 in septic patients | 7 days or less (may be discharged from critical care before day 7)
  Assess the concentration (e.g. umol/L) of circulating evolocumab and free (unbound by antibody) PCSK9 in evolocumab-treated patients with sepsis and compare to placebo controls.
Cmax of circulating evolocumab and circulating free PCSK9 in septic patients | 7 days or less (may be discharged from critical care before day 7)
  Assess the Cmax of circulating evolocumab and free (unbound by antibody) PCSK9 in evolocumab-treated patients with sepsis and compare to placebo controls.
Days alive | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in days alive over 28 days are associated with treatment arm.
Changes in 28-day mortality | 28 days
  Determine whether differences in mortality rates at 28 days exist between treatment arms.
Level of organ dysfunction | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in days free of organ dysfunction (cardiovascular, respiratory, renal, hematologic, and hepatic) over 28 days are associated with treatment arm.
Level of organ support | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in days free of organ support (vasopressor, ventilation and renal replacement therapy (RRT)) over 28 days are associated with treatment arm.
Changes in Vitals: lactate | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in plasma lactate levels (mmol/L) are associated with treatment arm.
Changes in Vitals: norepinephrine dose | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in norepinephrine levels (mcg/min) are associated with treatment arm.
Changes in Vitals: mean arterial pressure | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in mean arterial pressure levels (mm Hg) are associated with treatment arm.
Changes in Vitals: heart rate | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in heart rate (beats per minute) are associated with treatment arm.
Changes in Vitals: respiratory rate | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in respiratory rate (breaths per minute) are associated with treatment arm.
Changes in Vitals: temperature | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in temperature (degrees Celsius) are associated with treatment arm.
Changes in Vitals: fluid balance | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in fluid balance (Liters) are associated with treatment arm.
Changes in Vitals: urine output | 28 days or less (may be discharged from critical care before day 28)
  Determine if changes in urine output (Liters) are associated with treatment arm.
Safety outcomes: Number of treatment-related adverse events as ranked by severity | Day 1 to Day 90
  Monitor and count by category, and evaluate severity and seriousness of any adverse events related to the intervention that occurs in this critical and previously untested population.
Safety outcomes: changes in blood cell counts | 28 days or less (may be discharged from critical care before day 28)
  Document changes in blood cell counts (cells/ml) including white blood cells, red blood cells, and platelets, and determine whether clinically significant changes are associated with treatment.
Safety outcomes: changes in coagulation | 28 days or less (may be discharged from critical care before day 28)
  Document changes in coagulation of blood by measuring Prothrombin Time (PT) and Partial Thromboplastin Time (PTT). Both measurements determine time to clotting (in seconds) of different clotting factors and are then used to calculate International Normalized Ratio (INR) which helps monitor effects of blood thinning medication, and determine whether clinically significant changes are associated with treatment.
Safety outcomes: changes in blood analytes | 28 days or less (may be discharged from critical care before day 28)
  Document changes in concentration (e.g. umol/mL) of blood analytes, including hemoglobin, glucose, glycated hemoglobin, potassium, sodium, chloride, bicarbonate, creatinine, calcium, triponine, magnesium, aminotransferase, and alanine aminotransferase, and determine whether clinically significant changes are associated with treatment.
Safety outcomes: changes in urine density | 28 days or less (may be discharged from critical care before day 28)
  Document changes in urine specific gravity (density relative to water) and determine whether clinically significant changes are associated with treatment.
Safety outcomes: changes in urine pH | 28 days or less (may be discharged from critical care before day 28)
  Document changes in urine pH and determine whether clinically significant changes are associated with treatment.
Safety outcomes: changes in concentration of ketones in urine | 28 days or less (may be discharged from critical care before day 28)
  Document changes in concentration of ketones (e.g. umol/L) in the urine and determine whether clinically significant changes are associated with treatment.
Safety outcomes: document other urine abnormalities if required | 28 days or less (may be discharged from critical care before day 28)
  Document presence of blood, nitrites, bacteria, or urinary casts in the urine (yes or no) and determine whether clinically significant changes are associated with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Boyd, MD, Principal Investigator — University of British Columbia, Providence Health Care
Locations (3):
- Canada (3):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cirstea M, Walley KR, Russell JA, Brunham LR, Genga KR, Boyd JH. Decreased high-density lipoprotein cholesterol level is an early prognostic marker for organ dysfunction and death in patients with suspected sepsis. J Crit Care. 2017 Apr;38:289-294. doi: 10.1016/j.jcrc.2016.11.041. Epub 2016 Dec 7. PMID 28013095
- [Background] Roveran Genga K, Lo C, Cirstea M, Zhou G, Walley KR, Russell JA, Levin A, Boyd JH. Two-year follow-up of patients with septic shock presenting with low HDL: the effect upon acute kidney injury, death and estimated glomerular filtration rate. J Intern Med. 2017 May;281(5):518-529. doi: 10.1111/joim.12601. Epub 2017 Mar 19. PMID 28317295
- [Background] Levels JH, Abraham PR, van den Ende A, van Deventer SJ. Distribution and kinetics of lipoprotein-bound endotoxin. Infect Immun. 2001 May;69(5):2821-8. doi: 10.1128/IAI.69.5.2821-2828.2001. PMID 11292694
- [Background] Levels JH, Abraham PR, van Barreveld EP, Meijers JC, van Deventer SJ. Distribution and kinetics of lipoprotein-bound lipoteichoic acid. Infect Immun. 2003 Jun;71(6):3280-4. doi: 10.1128/IAI.71.6.3280-3284.2003. PMID 12761109
- [Background] Levels JH, Marquart JA, Abraham PR, van den Ende AE, Molhuizen HO, van Deventer SJ, Meijers JC. Lipopolysaccharide is transferred from high-density to low-density lipoproteins by lipopolysaccharide-binding protein and phospholipid transfer protein. Infect Immun. 2005 Apr;73(4):2321-6. doi: 10.1128/IAI.73.4.2321-2326.2005. PMID 15784577
- [Background] Topchiy E, Cirstea M, Kong HJ, Boyd JH, Wang Y, Russell JA, Walley KR. Lipopolysaccharide Is Cleared from the Circulation by Hepatocytes via the Low Density Lipoprotein Receptor. PLoS One. 2016 May 12;11(5):e0155030. doi: 10.1371/journal.pone.0155030. eCollection 2016. PMID 27171436
- [Background] Walley KR, Thain KR, Russell JA, Reilly MP, Meyer NJ, Ferguson JF, Christie JD, Nakada TA, Fjell CD, Thair SA, Cirstea MS, Boyd JH. PCSK9 is a critical regulator of the innate immune response and septic shock outcome. Sci Transl Med. 2014 Oct 15;6(258):258ra143. doi: 10.1126/scitranslmed.3008782. PMID 25320235
- [Background] Boyd JH, Fjell CD, Russell JA, Sirounis D, Cirstea MS, Walley KR. Increased Plasma PCSK9 Levels Are Associated with Reduced Endotoxin Clearance and the Development of Acute Organ Failures during Sepsis. J Innate Immun. 2016;8(2):211-20. doi: 10.1159/000442976. Epub 2016 Jan 13. PMID 26756586